CLINICAL TRIAL: NCT07152093
Title: Development of an Artificial Intelligence-Based Model for Predicting Difficult Intubation Using Video Laryngoscopic Images and Cormack-Lehane Classification
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Gizem Demir Şenoğlu, Principal Investigator, Assistant Professor of Anesthesiology and Reanimation, Düzce University Faculty of Medicine, Duzce University
Other Study IDs: 2025/183
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Difficult Airway Intubation
Keywords: Difficult Airway; Cormack-Lehane; Video Laryngoscopy; Artificial Intelligence; Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Normal Intubation Group: Intubations in patients assessed as Cormack-Lehane (CL) Class 1-2.
- Difficult Intubation Group: Intubations in patients evaluated as Cormack-Lehane Class 3-4.

SUMMARY:
This prospective observational study aims to develop an artificial intelligence model that can automatically determine the Cormack-Lehane classification from video laryngoscopy images in patients undergoing elective surgery. It also aims to predict the risk of difficult intubation based on this classification. The resulting data will evaluate the applicability of AI-supported decision support systems in clinical airway management.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years

Elective surgery

ASA I-II

No upper airway pathology

Exclusion Criteria:

* Known history of difficult intubation

Morbid obesity (BMI > 40)

Pregnancy

History of upper airway surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients undergoing elective surgery under general anesthesia at the operating rooms of Düzce University Medical Faculty Hospital. All patients will have their airways assessed using video laryngoscopy as part of routine anesthesia induction. Only patients without known upper airway pathology will be included.
  Patients will be prospectively and consecutively recruited. Video laryngoscopy images will be captured during intubation and used for machine learning analysis. The Cormack-Lehane grade will be independently confirmed by two experienced anesthesiologists. Patients will be classified into normal and difficult intubation groups.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Machine Learning Model in Predicting Difficult Intubation Based on Video Laryngoscopy Images | Immediately after data collection and model training
  The primary outcome is the classification accuracy of the machine learning algorithm in identifying difficult intubation cases (Cormack-Lehane grade 3-4) from video laryngoscopy images, compared with expert anesthesiologists' consensus. Accuracy will be reported as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Faculty of Medicine, Department of Anesthesiology and Reanimation, Düzce, Merkez, Turkey (Türkiye)